CLINICAL TRIAL: NCT01660776
Title: BMS_PD-L1_onco : Assessment of the PD-L1 Protein as a Biomarker in Oncology and Hematology
Acronym: BMS_PD-L1
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Roche Pharma AG (Industry); National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A01163-38; B111181-40 (Other: AFSSAPS); 11/32-821 (Other: CPP OUest V)
Record Dates: First submitted 2012-07-31; First posted 2012-08-09 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Diffuse Large B-cell Lymphoma; Hodgkin Lymphoma; Metastatic Breastcancer; Non-small Cell Lung Cancer
Keywords: diffuse large B-cell lymphoma (DLBCL); Hodgkin lymphoma; metastatic breast cancer.; non-small cell lung cancer
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomedical research on total blood at diagnosis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- DLBCL (diffuse large B-cell lymphoma): DLBCL (diffuse large B-cell lymphoma)
- Hodgkin's lymphoma: Hodgkin's lymphoma
- metastatic breast cancer: metastatic breast cancer or with lymph node involvement
- immune thrombocytopenia (ITP): immune thrombocytopenia (ITP)
- healthy volunteers: healthy volunteers
- non-small cell lung cancer: non-small cell lung cancer

SUMMARY:
Diffuse large B-cell lymphomas (DLBCLs) represent 25 to 30% of adult non-Hodgkin lymphomas in western countries. DLBCLs are aggressive cancer but potentially curable with multi-agent chemotherapy. Whereas R-CHOP regimen has led to a marked improvement in survival, this disease remains a biologically heterogeneous entity. New therapeutic strategies are required including identification of patients' subgroups with different prognostic.

This project is based on BMS_LyTrans and Goelams 075 clinical trial. A study of whole blood transcriptome in 75 DLBCL patients and in 87 controls showed that PD-L1 (CD274) gene was overexpressed in DLBCL patients. Preliminary results demonstrated that PD-L1 is detected in plasma of DLBCL patients with a significantly higher concentration than in controls. This protein was selected as a potential biomarker because of its established role in anti-tumoral immunity. Interaction between PD-L1 and its receptor PD-1 is known to inhibit activation of immune responses by inducing T-lymphocytes anergy and/or apoptosis. Moreover, a direct involvement of PD-L1 in the protection of cancer cells from lysis by activated T lymphocytes has been demonstrated. PD-L1 expression has been described in several solid tumours, including ovary cancer, breast cancer, colon cancer, renal cell carcinoma, non-small cell lung carcinoma and in hematological malignancies such as T-NHL, MM and Hodgkin's lymphoma. Furthermore the expression of PD-L1 by tumour cells is associated with poor prognosis. The blockade of PD-L1/PD-1 axis may represent a novel therapeutic approach in aggressive cancers. These first results incite to identify the cells releasing soluble PD-L1 and to investigate its role in the anti-tumoral immunity in DLBCL patients.

The aim of this study is to identify cells producing soluble PD-L1 in DLBCL patients at diagnosis in comparison to others tumours known to express PD-L1 (metastatic breast cancer, Hodgkin's lymphoma, non-small cell lung cancer).

DETAILED DESCRIPTION:
Secondary purposes are :

* To confirm the presence of plasma soluble form of PD-L1 in others malignancies
* To study surface expression of PD-L1 on circulating tumour cells with multiparameter fow cytometry and Veridex® technology in DLBCL and metastatic breast cancer patients
* To study surface expression of PD-L1 on circulating endothelial cells in DLBCL, Hodgkin lymphoma and metastatic breast cancer patients (subpart ended in late 2012)
* To study surface expression of PD-L1 on different types of leukocytes (monocytes, B and T lymphocytes)
* To separate circulating tumour cells expressing PD-L1 by immunomagnetic or Cell-sorting method
* To develop ELISPOT technique to study the release of soluble PD-L1 in culture supernatants of selected cells (subpart ended mid 2013)
* to evaluate the correlation between the expression of PD-L1 in the plasma and *) the expression of PD-L1 in the tumor, **) the expression of PD-L1 and other molecules in the bronchoalveolar liquid (whenever available from routine) in non-small cell lung cancer
* to evaluate the response to treatment according to plasma PD-L1 expression in non-small cell lung cancer
* to evaluate the susceptibility to develop a disease according to the single nucleotide polymorphisms of the PD-L1 gene in DLBCL and non-small cell lung cancer
* Constitution of the different cohorts and collection of samples Main cohort : de novo DLBCL at diagnosis Secondary cohorts: Hodgkin's lymphoma, metastatic breast cancer, non small cell lung cancer Control cohorts : healthy volunteers (blood donors), patients with immune thrombocytopenia (ITP)
* Quantification of plasma soluble PD-L1 in the different cohorts

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria :

* Age ≥ 18 years and ≤ 75 years,
* Life expectancy more than 4 months
* Signed informed consent obtained
* Social security affiliation is mandatory
* Non previously treated (even by corticotherapy),
* HIV negative, HBs negative, HCV negative

Inclusion criteria for DLBCL patients :

* A biopsy proven diagnosis of de novo DLBCL according to the current WHO criteria,
* Immunohistochemistry for GCB/nonGC classification according to Hans' algorithm
* Patients with advanced-stage disease defined as Ann Arbor stages III or IV, or stages I or II with bulky disease (>7cm)

Inclusion criteria for non-small cell lung cancer patients :

* A biopsy proven diagnosis of de novo non-small cell lung cancer (all stages) according to the current WHO criteria

Inclusion criteria for Hodgkin's lymphoma patients :

* A biopsy proven diagnosis of Hodgkin's lymphoma according to the current WHO criteria

Inclusion criteria for metastatic breast cancer or with lymph node involvement :

* A biopsy proven diagnosis infiltrating lobular or ductal breast carcinoma
* with lymph node involvement or metastasis

Inclusion criteria for patients with immune thrombocytopenia (ITP) :

* Primary ITP was defined by the IWG as a platelet count less than 100 G/L in the absence of other causes or disorders that may be associated with thrombocytopenia.
* Bone marrow examination excluding a central aetiology of thrombocytopenia

Inclusion criteria for healthy volunteers :

- Inclusion criteria for blood donation according to the Etablissement Français du Sang (EFS) criteria

Exclusion Criteria:

General non-inclusion criteria :

* Age < 18 years et > 75 years,
* Pregnant women,
* Person legally involved in a case
* No social security affiliation
* Signed informed consent not obtained,
* Preliminary treatment (even corticoid treatment).
* HIV positive, HBs positive, HCV positive

Non-inclusion criteria for DLBCL patients :

* Lymphoma other than DLBCL,
* Transformation of a low grade lymphoma to a high grade lymphoma (DLBCL),
* Extranodal marginal zone lymphoma of MALT lymphoma,
* Post-transplant lymphoproliferative disorders,
* Lymphoblastic lymphoma,
* Burkitt's lymphoma,
* Carcinoma or history of carcinoma except in situ cervical carcinoma.

Non-inclusion criteria for non-small cell lung cancer patients : None

Non-inclusion criteria for Hodgkin patients :

- Non Hodgkin's lymphoma

Non-inclusion criteria for metastatic breast cancer or with lymph node involvement :

* Carcinoma other than infiltrating lobular or ductal breast carcinoma
* Chemotherapy in 30 days preceding the inclusion
* Hormonotherapy in 7 days preceding the inclusion
* Carcinoma or history of carcinoma except in situ cervical carcinoma.
* Hemoglobin level < 10g/dl

Non-inclusion criteria for patients with immune thrombocytopenia (ITP) :

- Central aetiology of the thrombocytopenia

Non-inclusion criteria for healthy volunteers :

- Exclusion criteria for blood donation according to the Etablissement Français du Sang (EFS) criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of DLBCL patients : 40 Number of non-small cell lung cancer patients : 100 Number of Hodgkin patients : 20 Number of metastatic breast cancer patients : 20 Number of healthy volunteers : 140 Number of patients with immune thrombocytopenia (ITP) : 5
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Description of one or several blood cell types producing soluble PD-L1 in DLBCL, metastatic breast cancer, Hodgkin's lymphoma and non-small cell lung cancer | 4 years
  Description of one or several blood cell types producing soluble PD-L1 in DLBCL, metastatic breast cancer, Hodgkin's lymphoma and non-small cell lung cancer

SECONDARY OUTCOMES:
Analysis of PD-L1 membrane protein expression on circulating tumor cells by multiparameter flow cytometry and Veridex® in DLBCL and metastatic breast cancer, and bone marrow tumor cells by flow cytometry in DLBCL | 4 years
  Analysis of PD-L1 membrane protein expression on circulating tumor cells by multiparameter flow cytometry and Veridex® in DLBCL and metastatic breast cancer, and bone marrow tumor cells by flow cytometry in DLBCL
Analysis of PD-L1 membrane protein expression on circulating endothelial cells with the Veridex® technology in DLBCL, Hodgkin's lymphoma and metastatic breast cancer (subpart ended in late 2012) | 4 years
  Analysis of PD-L1 membrane protein expression on circulating endothelial cells with the Veridex® technology in DLBCL, Hodgkin's lymphoma and metastatic breast cancer (subpart ended in late 2012)
Analysis of PD-L1 membrane protein expression on monocytes, B and T lymphocytes in all cohorts | 4 years
  Analysis of PD-L1 membrane protein expression on monocytes, B and T lymphocytes in all cohorts
Development of an ELISPOT technique to detect soluble PD-L1 in the supernatants of sorted primary cells (subpart ended mid 2013) | 4 years
  Development of an ELISPOT technique to detect soluble PD-L1 in the supernatants of sorted primary cells (subpart ended mid 2013)
Evaluation of the techniques (by immunomagnetic or cell-sorting) used to separate circulating tumor cells expressing PD-L1 | 4 years
  Evaluation of the techniques (by immunomagnetic or cell-sorting) used to separate circulating tumor cells expressing PD-L1
Correlation between the PD-L1 expression *) in the plasma, **) in the tumor and ***) in the bronchoalveolar liquid in non-small cell lung cancer | 4 years
  Correlation between the PD-L1 expression *) in the plasma, **) in the tumor and ***) in the bronchoalveolar liquid in non-small cell lung cancer
Evaluation of the response to treatment according to soluble PD-L1 expression in non-small cell lung cancer | 4 years
  Evaluation of the response to treatment according to soluble PD-L1 expression in non-small cell lung cancer
Evaluation of the susceptibility to develop a disease according to PD-L1 gene SNP in DLBCL and non-small cell lung cancer | 4 years
  Evaluation of the susceptibility to develop a disease according to PD-L1 gene SNP in DLBCL and non-small cell lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Fest, MD, Principal Investigator — Rennes University Hospital
Locations (4):
- France (4):
  - Rennes EFS, Rennes, Brittanny
  - Rennes University Hospital, Rennes, Brittanny
  - Institut Paoli Calmette, Marseille
  - Montpellier University Hospital, Montpellier